CLINICAL TRIAL: NCT02426554
Title: Dietary Supplementation of of DHA, Vitamin D3 and Uridine in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Technical University of Denmark (Other); Helene Elsass Center, Denmark. (Unknown)
Responsible Party: Principal Investigator, Solvejg Hansen, Cand Scient Human Physiology, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: Braindrop
Record Dates: First submitted 2015-04-16; First posted 2015-04-27 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-08

CONDITIONS: Children

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Active Comparator)
  Interventions: Dietary Supplement: DDU-supplement
- Group 2 (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo supplement

INTERVENTIONS:
Dietary Supplement: DDU-supplement — DDU: Vitamin D, DHA, Uridine
  Arms: Group 1
Dietary Supplement: Placebo supplement
  Arms: Group 2

SUMMARY:
The feasibility of combining a motor and cognitive exercise program with dietary supplementation (DDU: Vitamin D, DHA and Uridine or Placebo) is tested in a smaller group of prepubescent children.

ELIGIBILITY:
Inclusion Criteria:

- age 8 to 11 yrs.

Exclusion Criteria:

* history of neurological or psychiatric disorders.

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2011-01; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Compliance to cognitive and motor training program (Move It To Improve It: MiTii) | 6 weeks
  Internet based program with evaluation of numbers of training sessions. At least 14 training sessions out of 18 should be completed.
Dietary compliance | 6 weeks
  Supplement was provided to the children and ingestion was registered by the parents.

CONTACTS AND LOCATIONS:
Overall Officials: Jens Bo Nielsen, Professor, Study Director — NEXS

REFERENCES:
- [Derived] Hansen SL, Ritterband-Rosenbaum A, Voigt CB, Hellgren LI, Sorensen AM, Jacobsen C, Greve LZ, Jorgensen KD, Bilde PE, Kiens B, Nielsen JB. Supplementation of docosahexaenoic acid (DHA), vitamin D3 and uridine in combination with six weeks of cognitive and motor training in prepubescent children: a pilot study. BMC Nutr. 2017 Apr 17;3:37. doi: 10.1186/s40795-017-0155-1. eCollection 2017. PMID 32153817